CLINICAL TRIAL: NCT04546490
Title: Effects of Pressure Release and Ischemic Pressure of Myofascial Trigger Points on Mechanical Neck Pain. A Crossover, Controlled and Randomized Clinical Trial
Brief Title: Effects of Release and Ischemic Pressure of Trigger Points on Neck Pain. A Crossover, Controlled and Randomized Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Iván Batuecas Sánchez, Máster Universitario en Cuidados de Salud, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C.I. 20/090-E
Record Dates: First submitted 2020-08-20; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Myofascial Trigger Point Pain; Myofascial Pain; Myofascial Pain Syndrome; Neck Pain
Keywords: Upper Trapezius Muscle; Manual therapy; Pressure Release Technique; Ischemic Pressure Technique
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain

STUDY DESIGN:
Intervention Model Description: Patients, aged 18-50 years with mechanical neck pain for at least the last month, will be randomly divided into three groups: one will be given Pressure Release technique, another Ischemic Pressure technique, and a last one will be assigned as a control group.
  They will be crosslinked after the first treatment. The variables will be evaluated before and immediately after treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know to which group they have been assigned in each of the interventions Participants will be assigned an individual code by which the outcome assessor will not be able to know what treatment(s) each individual received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pressure release (Experimental): It will be applied with the patient in a supine position. The therapist will clamp his first and second fingers over the Myofascial Trigger Point located on the upper trapezium, it will be marked previously. The pressure will increase as the therapist perceives a reduction in the resistance offered by the soft tissue under his finger within a period of 90 seconds.
  Interventions: Other: Pressure Release technique; Other: Ischemic pressure technique
- Ischemic pressure (Experimental): Patient in supine position, the therapist performs pressure with first and second finger in PGM marked previously, this is performed until the patient tolerance, when the patient refers a decrease in pain or have a correct adaptation to the perceived pain increase the pressure to a new painful barrier. Repeat the process for 90 seconds.
  Interventions: Other: Pressure Release technique; Other: Ischemic pressure technique
- Control Group (No Intervention): Patient in supine position on the stretcher, the therapist performs a clamp with the first and second finger on the upper trapezius muscle without making any pressure on it during 90 seconds

INTERVENTIONS:
Other: Pressure Release technique — Manual therapy technique used by the treatment of Myofsacial Trigger points. The therapist will apply it with the first and second finger on the previously marked Myofascial Trigger Point and increasing the pressure as he perceives a reduction in the resistance offered by the soft tissue under the finger
  Arms: Ischemic pressure; Pressure release
Other: Ischemic pressure technique — Manual therapy technique by making pressure in Myofascial Trigger Point. The therapist will apply it with the first and second finger on the previously marked Myofascial Trigger Point. This is performed until the patient's tolerance, when he refers a decrease in pain or have a correct adaptation to the perceived pain increase the pressure to a new painful barrier.
  Arms: Ischemic pressure; Pressure release

SUMMARY:
The aim of the study is to compare two manual therapy techniques. By testing if the Pressure Release of Myofascial Trigger Points technique (PRM) is more effective in treating Myofascial Trigger Points present in the upper trapezius muscle of patients with mechanical cervical pain. This will be compared mainly with another manual therapy technique that presents evidences such as Ischemic Pressure technique (IP), and a control group, through the evaluation of the Visual Analogical Scale (VAS), the Threshold of Pain at Pressure (TPP) and the Northwick Park Questionnaire (NPC) of neck disability, spanish version.

DETAILED DESCRIPTION:
The present pilot study is proposed as a crossover, controlled and randomized clinical trial, with blinded evaluation of response variables.

The aim of the study is to test whether the Pressure Release of Myofascial Trigger Points technique(PRM) is effective in treating Myofascial Trigger Points present in the upper trapezius muscle of patients with mechanical cervical pain. This will be compared mainly with another manual technique that presents more evidence such as Ischemic Pressure (IP), through the evaluation of the Visual Analogical Scale (VAS), the Threshold of Pain at Pressure (TPP) and the Northwick Park Questionnaire (NPC) of neck disability, Spanish version.

The patients, with a minimum sample for the pilot study of 30 subjects, of working age (18-50 years) with mechanical neck pain for at least the last month, will be recruited from the clinic "Fisioterapia Los Molinos" in the town of Getafe, the same place where the treatment will be carried out.

They will be randomly divided into three groups: one will be given Pressure Release of Myofascial Trigger Points technique (PRM), another Ischemic Pressure technique (IP), and a last one will be assigned as a control group. In compliance with the corresponding ethical criteria, the three groups will be subjected to random crossover so that no patient is left untreated. Visual Analogical Scale (VAS), Threshold of Pain at Pressure (TPP) and Northwick Park Questionnaire (NPC) of neck disability (spanish version), will be evaluated before and immediately after treatment.

Statistical analysis will be performed by IBM SPSS v22.0 program or a later version, verifying that the sample meets the criteria of normality and homogeneity and comparing the results of the variables through an ANOVA Analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* patients with neck pain in the last month

Exclusion Criteria:

* Patients with recent surgeries of the upper quadrant or spine.
* Patients who are currently undergoing pharmacological or physiotherapeutic treatment.
* Patients who have suffered a recent traffic accident or other type of trauma
* Patients who are in the gestation period.
* Patients who have malignant neoplasms.
* Patients who do not sign the informed consent, do not understand the Spanish language or any other circumstance that would prevent their participation in this research will also be discarded
* Patients with no palpable active or latent myofascial trigger points in the upper trapezius muscle

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Before the intervention
  Place a mark in a chart according to the state of pain you are in at the moment, taking into account that the left extreme is the absence of pain and the opposite is the worst pain you may suffer
Visual Analog Scale | immediately after the intervention
  Place a mark in a chart according to the state of pain you are in at the moment, taking into account that the left extreme is the absence of pain and the opposite is the worst pain you may suffer
Pain Threshold at Pressure | Before the intervention
  Evaluated with a pressure algometer. It will be assessed with the subject in a comfortable position, back supported by the backrest, feet on the floor and arms relaxed. The algometer will be placed perpendicular to the previously marked Miofascial Trigger Point. Once it is in place, the pressure should be increased one kilogram by second until the patient begins to feel discomfort.
  At this point the application will be stopped. Three measurements were made and the average will be calculated. Measured by Kilograms per square centimeter
Pain Threshold at Pressure | immediately after the intervention
  Evaluated with a pressure algometer. It will be assessed with the subject in a comfortable position, back supported by the backrest, feet on the floor and arms relaxed. The algometer will be placed perpendicular to the previously marked Miofascial Trigger Point. Once it is in place, the pressure should be increased one kilogram by second until the patient begins to feel discomfort.
  At this point the application will be stopped. Three measurements were made and the average will be calculated. Measured by Kilograms per square centimeter
Northwick Park Questionary (Spanish Modified Version) for Cervical Spine disability | Before the intervention
  The questionnaire consists of nine questions related to pain intensity, sleep, weight load, leisure and social activities, work and driving. Each one of them presents five possible answers graduated from 0 to 4, where 0 represents the absence of disability and 4 the maximum degree of disability.
Northwick Park Questionary (Spanish Modified Version) for Cervical Spine disability | immediately after the intervention
  The questionnaire consists of nine questions related to pain intensity, sleep, weight load, leisure and social activities, work and driving. Each one of them presents five possible answers graduated from 0 to 4, where 0 represents the absence of disability and 4 the maximum degree of disability.

SECONDARY OUTCOMES:
Height | Before the first intervention
  Height of the subject
Weight | Before the first intervention
  Weight of the subject
Age | Before the first intervention
  Age of the subject
Sex | Before the first intervention
  Sex of the subject
Working Status | Before the first intervention
  Working status of the subject

CONTACTS AND LOCATIONS:
Locations (1):
- Fisioterapia Los Molinos, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided